CLINICAL TRIAL: NCT02989142
Title: Inter-pregnAncy Coaching for a Healthy fuTure
Acronym: inter-act
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: KU Leuven (Other)
Collaborators: Universiteit Antwerpen (Other); UC Leuven-Limburg (Unknown)
Responsible Party: Principal Investigator, dr. Annick Bogaerts, Prof. dr., KU Leuven
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: T005116N
Record Dates: First submitted 2016-08-29; First posted 2016-12-12 (Estimated); Last update posted 2017-06-12 (Actual); Status verified 2017-06

CONDITIONS: Obesity; Pregnancy
Keywords: interpregnancy; pregnancy-induced hypertension; gestational diabetes mellitus; caesarean section; large-for-gestational-age
MeSH Terms: conditions — Obesity; Hypertension, Pregnancy-Induced; Diabetes, Gestational

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control arm (No Intervention): No intervention
- INTER-ACT arm (Experimental): Four pre-conception coaching sessions : postpartum week 6, week 8, week 12, 6 months.
  Three pregnancy coaching sessions: at the time of the planned ultrasound scans.
  Interventions: Behavioral: INTER-ACT

INTERVENTIONS:
Behavioral: INTER-ACT — Pre-conception coaching sessions: We encourage less motivated women to participate to the trial by collaborating with Kind & Gezin from the very beginning, as most timepoints of the counselling sessions coincide with the time points of the Kind&Gezin vaccine scheme (postpartum week 6, week 8, week 12, 6 months). We will organize the coaching in a "mother and baby friendly" community-based setting or in the hospitals, as preferred by the mothers.
  Pregnancy coaching sessions: take place in hospital, at the time of the three planned ultrasound scans.
  By consequence, the applied methodology can be applied as such at the moment of global utilisation in Flanders.
  Arms: INTER-ACT arm

SUMMARY:
The project focuses on prevention of major pregnancy and birth related complications : pregnancy-induced hypertension (PIH), gestational diabetes mellitus (GDM), caesarean section (CS), and large-for-gestational-age (LGA), i.e. the birth weight of the baby exceeds the 90% percentile of birth weights for the specific pregnancy duration.

The investigators focus on the pre-conception period, i.e. the pre-conception period of the 2nd pregnancy in women with an excessive weight gain during their 1st pregnancy, aiming to decrease the complications rate in their 2nd pregnancy.

Women with an excessive gestational weight gain have obtained the extra weight during a rather short period of time, e.g. 20 kilos in the last 4 or 5 months of their pregnancy. This characteristic distinguishes the target group from the general population with overweight/obesity, in whom the extra weight was acquired during many years and independent from a pregnancy, making a behaviour change more complex.

The coaching intervention combines face-to-face counselling with the use of a mobile App connected to medical devices (scale and pedometer). The app monitors important indicators (weight, eating behaviour, physical activity, mental wellbeing), provides coaching through established behavioral change techniques, and is specifically tailored for women with excessive weight gain during the previous pregnancy.

The goal is to decrease the rate of pregnancy and birth-related adverse outcomes in the next pregnancy by a healthy life style, starting shortly after their 1st delivery and sustained during the next pregnancy.

DETAILED DESCRIPTION:
The aim is to decrease the prevalence of pregnancy and birth-related complications (pregnancy-induced hypertension (PIH), gestational diabetes mellitus (GDM), caesarean section (CS), and large-for-gestational-age babies (LGA)). These complications occur in 26% of pregnancies with normal start BMI and adequate weight gain, in 34% in normal start BMI but excessive gestational weight gain and in up to 66% in obese class III (BMI≥40kg/m²) combined with excessive gestational weight gain. Moreover, as the prevalence of maternal obesity continues to rise, increasing numbers of children are exposed to an 'obesogenic intrauterine environment'. Obesity in pregnancy has therefore the potential to result in an 'intergenerational cycle' of obesity through in utero programming.

The investigators focus on women with excessive weight gain during their 1st pregnancy as currently, half of them do not return to their pre-pregnancy weight before the next pregnancy. This results in a complication rate as high as 42% (PIH, GDM, CS, LGA). The investigators target a healthy BMI at start of pregnancy by intervening during the pre-conception period- and an adequate weight gain during pregnancy by intervening during pregnancy in these women. The intervention will be evaluated in a randomized controlled trial including 1,100 women.

The proposed intervention combines face-to-face coaching with the use of a mobile App (so-called 'inter-act' app) connected to medical devices (scale and pedometer). The app monitors women's weight, eating behaviour, physical activity, mental wellbeing, and provides continuously coaching through positive behavioral change techniques. The 'inter-act' App covers after the 1st delivery breast-feeding support, while during pregnancy, the gestational weight gain guidelines of the Institute of Medicine (IOM) are included.

Drop out of less motivated women is avoided as the time points of the four pre-conception coaching sessions coincide with the existing postnatal follow-up visits for neonates (Governmental vaccination scheme through the organisation " Kind & Gezin"), and the three pregnancy coaching sessions coincide with the three routine ultrasound scans during normal pregnancy (KCE Guidelines).

Each year, there are 8,900 singleton pregnancies in Flanders in whom the mother had excessive gestational weight gain in the prior pregnancy. The current rate of at least one of the four major pregnancy and birth-related complications (PIH, GDM, CS, LGA) in the 8,900 pregnancies is 42%. If the complications rate reduces with 1/4, this involves more than 900 pregnancies, and reduces costs related to caesarean sections, gestational diabetes, obesity in mother & child.

ELIGIBILITY:
Inclusion Criteria:

* Excessive weight gain during their previous pregnancy (above the IOM recommendations)
* Child wish for having a next pregnancy
* Women aged 18 years or more
* Sufficient fluent in Dutch language
* Able to give written informed consent
* Able to use a smartphone. If the women do not have a smartphone because of socio-economic reasons, a smartphone is at her disposal for the whole duration of the intervention, in order to be able to use Apps connected with a Bluetooth pedometer and balance scale.

Exclusion Criteria:

* Requirement for (complex) diets
* History of or a plan for bariatric surgery
* Underlying or chronic disorders (e.g. diabetes, thyroid disease, renal diseases)
* Significant psychiatric disorder
* Previous still birth

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1100 (Estimated)
Dates: Start 2017-04-01 (Actual); Primary Completion 2020-03 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
prevalence of participants with at least one of the following four complications: pregnancy-induced hypertension, gestational diabetes mellitus, caesarean section, large-for-gestational age baby | at the time of delivery 2nd pregnancy (max pregnancy duration 44 weeks)
  The existence of pregnancy-induced hypertension and gestational diabetes mellitus are assessed during pregnancy. Whether the 2nd pregnancy results in a caesarean section and large-for-gestational-age baby will be known at the time of delivery 2nd pregnancy. Therefore, the primary outcome of prevalence of participants with pregnancy and birth-related complications is assessed at the time of delivery 2nd pregnancy.

SECONDARY OUTCOMES:
Drop out | at 6 months, at 12 months, at 18 months .... till delivery 2nd pregnancy
  Drop-out rate and reason for drop-out
Rate of women who returned to their pre-pregnancy weight | at 6 months, at 12 months, at 18 months .... till delivery 2nd pregnancy
Distribution underweight, normal weight, overweight, obese BMI | at 6 months, at 12 months, at 18 months .... till delivery 2nd pregnancy
Body composition | at 6 months, at 12 months, at 18 months .... till delivery 2nd pregnancy
  Body composition measured by bio-electrical impedance analysis to estimate fat mass, fat free mass and muscle mass.
Skin fold measurements | at 6 months, at 12 months, at 18 months .... till delivery 2nd pregnancy
  Skin fold measurements or determining body fat composition by use of a skinfold calliper.
Breast feeding behaviour | at 6 months, at 12 months, at 18 months .... till delivery 2nd pregnancy
  Breast feeding (BF) habits are assessed by a structured questionnaire on breastfeeding practice. The questionnaire consists of eleven questions in Dutch, which investigates intention to BF, initiation to BF, exclusive BF, combination of bottle-feeding and BF and motives to cease BF.
Food intake | at 6 months, at 12 months, at 18 months .... till delivery 2nd pregnancy
  food intake is measured by a Food Frequency Questionnaire: frequency of food intake (per day, per week or per month) and portion size (in gram or millilitre).
Physical activity | at 6 months, at 12 months, at 18 months .... till delivery 2nd pregnancy
  Physical activity is measured using International Physical Activity Questionnaire (IPAQ), long version.
Life style behaviour | at 6 months, at 12 months, at 18 months .... till delivery 2nd pregnancy
  Life style behaviour: whether the mother is following a diet, smoking, sleep duration and quality of sleep, alcohol use (questionnaire).
Anxiety | at 6 months, at 12 months, at 18 months .... till delivery 2nd pregnancy
  Anxiety symptoms are measured with the Trait Anxiety Inventory (TAI).
Depression | at 6 months, at 12 months, at 18 months .... till delivery 2nd pregnancy
  Levels of depression are measured with the reliable and valid 10-item Edinburgh Postnatal Depression Scale (PDS).
rate of patients with excessive gestational weight gain during their 2nd pregnancy. | at the time of delivery 2nd pregnancy (max pregnancy duration 44 weeks)
Rate of preterm/term pregnancies | at the time of delivery 2nd pregnancy (max pregnancy duration 44 weeks)
Cost-effectiveness of the intervention | at the time of delivery 2nd pregnancy (max pregnancy duration 44 weeks)
  Costs related to these complications:
  1. caesarean section costs 4,013€ compared to 2,909€ for a vaginal delivery, resulting in a 4,013-2,909= 1,104€ additional cost per caesarean section (Onafhankelijke Ziekenfondsen, 2012).
  2. Gestational diabetes has an additional cost 820 € (Danyliv et al., IADPSG 2014, Gestational Diabetes and health care cost).
  3. There is also the impact of gestational diabetes on the baby. Intrauterine exposure through gestational diabetes predisposes the off-spring to diabetes: yearly cost for diabetes around 5,800€ (American Diabetes Association).
  4. Obesity: yearly additional direct medical cost for obesity approximately 3000 € per person due to increased contacts with health care providers and hospitalisation costs (De Jonghe E and Annemans L, 2009).
  The costs of the coaching sessions are based on the official nomenclature of midwives (RIZIV - Rijksinstituut voor ziekte- en invaliditeitsverzekering, Belgian institute)
Number of women who gave at least 6 months breast feeding | at 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Roland Devlieger, PhD, MD, Study Chair — Katholieke Universiteit Leuven, Department of Development and Regeneration
Locations (6):
- Belgium (6):
  - UZA, Antwerp
  - Ziekenhuizen GasthuisZusters Antwerpen (GZA), Antwerp
  - Ziekenhuis Oost-Limburg (ZOL), Genk
  - Jessa ziekenhuis, Hasselt
  - Sint-Franciskusziekenhuis, Heusden
  - UZ Leuven, Leuven

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Van Uytsel H, Ameye L, Devlieger R, Bijlholt M, Van der Gucht K, Jacquemyn Y, Bogaerts A. Effect of the INTER-ACT lifestyle intervention on maternal mental health during the first year after childbirth: A randomized controlled trial. PLoS One. 2023 Jul 28;18(7):e0284770. doi: 10.1371/journal.pone.0284770. eCollection 2023. PMID 37506163
- [Derived] Van Uytsel H, Bijlholt M, Devlieger R, Ameye L, Jochems L, van Holsbeke C, Schreurs A, Catry V, Bogaerts A. Effect of the e-health supported INTER-ACT lifestyle intervention on postpartum weight retention and body composition, and associations with lifestyle behavior: A randomized controlled trial. Prev Med. 2022 Nov;164:107321. doi: 10.1016/j.ypmed.2022.107321. Epub 2022 Oct 27. PMID 36309119
- [Derived] Bijlholt M, Ameye L, Van Uytsel H, Devlieger R, Bogaerts A. The INTER-ACT E-Health Supported Lifestyle Intervention Improves Postpartum Food Intake and Eating Behavior, but Not Physical Activity and Sedentary Behavior-A Randomized Controlled Trial. Nutrients. 2021 Apr 14;13(4):1287. doi: 10.3390/nu13041287. PMID 33919758
- [Derived] Bogaerts A, Ameye L, Bijlholt M, Amuli K, Heynickx D, Devlieger R. INTER-ACT: prevention of pregnancy complications through an e-health driven interpregnancy lifestyle intervention - study protocol of a multicentre randomised controlled trial. BMC Pregnancy Childbirth. 2017 May 26;17(1):154. doi: 10.1186/s12884-017-1336-2. PMID 28549455